CLINICAL TRIAL: NCT06547203
Title: Negative Ultraselection of Patients With RAS/BRAF Wild-type Refractory Right-Sided Metastatic Colorectal Cancer Receiving Cetuximab in Combination With Toripalimab and Irinotecan: A Phase II, Single-arm Study
Brief Title: Cetuximab, Irinotecan, Toripalimab in RAS/BRAF Wild-type Ultraselected Right-sided Colorectal Cancer Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITRUS
Record Dates: First submitted 2024-07-18; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastatic colorectal cancer; RAS/BRAF wild type; Right-sided; Cetuximab; PD-1 inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; toripalimab; Irinotecan

STUDY DESIGN:
Intervention Model Description: To investigate the objective response rate (ORR) of cetuximab combined with toripalimab and irinotecan in right-sided mCRC patients with negative ultraselected RAS/BRAF wild-type who have progressed after previous treatments with bevacizumab, irinotecan, oxaliplatin, and 5-fluorouracil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cetuimab plus toripalimab and irinotecan (Experimental): Single Arm study, with patients receiving:
  Cetuximab: 500 mg/m², intravenous infusion, once every 2 weeks. Toripalimab: 3 mg/kg, intravenous infusion, once every 2 weeks. Irinotecan: 150 mg/m², intravenous infusion, once every 2 weeks.
  Patients will continue treatment until any of the following conditions occur: the researcher determines there is no longer a clinical benefit, intolerable toxicity occurs, a new anti-tumor treatment is initiated, withdrawal of informed consent, loss to follow-up, death, or other conditions specified in the protocol requiring termination of treatment.
  Interventions: Drug: Cetuximab; Drug: Toripalimab; Drug: Irinotecan

INTERVENTIONS:
Drug: Cetuximab — Cetuximab: 500 mg/m², intravenous infusion, once every 2 weeks
  Other Names: Erbitux
Drug: Toripalimab — Toripalimab: 3 mg/kg, intravenous infusion, once every 2 weeks.
  Other Names: Loqtorzi
Drug: Irinotecan — Irinotecan: 150 mg/m², intravenous infusion, once every 2 weeks.
  Other Names: CPT-11

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of cetuximab combined with PD-1 inhibitor and irinotecan in negative ultraselection RAS/BRAF wild-type refractory right-sided metastatic colorectal cancer.

DETAILED DESCRIPTION:
The present study focuses on exploring the effectiveness and safety of cetuximab combined with a PD-1 inhibitor and irinotecan in treating refractory, right-sided metastatic colorectal cancer (mCRC) patients who are negative ultraselected for RAS/BRAF mutations. Colorectal cancer ranks among the most prevalent digestive malignancies globally, with right-sided mCRC generally exhibiting poorer outcomes than left-sided cases. Current treatment guidelines vary based on genetic mutations and tumor location, recommending cetuximab for left-sided RAS/BRAF wild-type mCRC and alternative therapies for right-sided or mutated cases. Despite limited clinical data on EGFR inhibitors for right-sided mCRC, retrospective analyses suggest varying efficacy outcomes. The study aims to address these gaps by investigating cetuximab and PD-1 inhibitor combination therapy in this specific patient population, potentially enhancing treatment options for refractory mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma.
* Primary tumor located in the right colon.
* Metastatic disease with at least one measurable lesion according to RECIST v1.1 criteria.
* Histologically tested as RAS/BRAF V600E wild-type and negative ultraselected for mutations including: RAS/BRAF V600E/PIK3CA/PTEN/EGFR (ECD), HER2 and MET amplification, and ALK/RET/NTRK1 gene fusions.
* Patients who have progressed after previous treatments including bevacizumab, irinotecan, oxaliplatin, and 5-fluorouracil, with tumor progression occurring during or within 3 months after irinotecan treatment.
* No prior treatment with anti-EGFR or PD-1 antibodies.
* Normal hematological function (platelets >90×10^9/L; white blood cells >3×10^9/L; neutrophils >1.5×10^9/L).
* Serum bilirubin ≤1.5 times the upper limit of normal (ULN), transaminases ≤5 times ULN.
* No ascites, normal coagulation function, albumin ≥35 g/L.
* Liver function classified as Child-Pugh grade A.
* Serum creatinine less than ULN, or calculated creatinine clearance >50 ml/min (using the Cockcroft-Gault formula).
* At least one measurable lesion according to RECIST v1.1 criteria.
* ECOG performance status of 0-2.
* Expected survival >3 months.
* Signed written informed consent.
* Willing and able to undergo follow-up until death or study completion or termination.

Exclusion Criteria:

* Severe arterial thrombosis or ascites.
* Bleeding tendencies or coagulation disorders.
* Hypertensive crisis or hypertensive encephalopathy.
* Severe uncontrolled systemic complications such as infections or diabetes.
* Clinically significant cardiovascular diseases such as cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), uncontrolled hypertension despite appropriate medication, unstable angina, congestive heart failure (NYHA grade 2-4), or arrhythmias requiring medication.
* History of or physical examination showing central nervous system diseases (e.g., primary brain tumor, uncontrolled epilepsy, any history of brain metastasis or stroke).
* Other malignancies within the past 5 years (except for basal cell carcinoma of the skin after curative surgery and/or carcinoma in situ of the cervix).
* Use of immunosuppressive drugs within 1 week before treatment, excluding nasal, inhaled, or other topical steroids or physiological doses of systemic steroids (i.e., not exceeding 10 mg/day of prednisone or an equivalent dose of other steroids) or steroids used to prevent contrast agent allergies.
* Steroid-dependent interstitial lung disease.
* Known active autoimmune disease requiring symptomatic treatment or history of such disease within the past 2 years. Patients with vitiligo, psoriasis, alopecia, or -Graves' disease not requiring systemic treatment within the past 2 years, hypothyroidism requiring only thyroid hormone replacement, and type I diabetes requiring only insulin replacement can be enrolled.
* Known history of primary immunodeficiency.
* Known active tuberculosis.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Receipt of any investigational drug treatment within the last 28 days before the study.
* Allergy to any drugs in the study.
* Pregnant or breastfeeding women.
* Women of childbearing potential (within 2 years of last menstruation) or men capable of fathering a child who are not using or refuse to use effective non-hormonal contraceptive methods (e.g., intrauterine device, barrier method combined with spermicide, or sterilization).
* Inability or unwillingness to comply with the study protocol.
* Presence of any other disease, functional impairment caused by metastatic lesions, or suspicious conditions found during a physical examination indicating a contraindication to the study drugs or high risk for treatment-related complications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Assessed after every 4 cycles (each cycle is 14 days) for up to 24 months
  The proportion of patients who have achieved partial response (PR) plus complete response (CR), as assessed by the investigator using RECIST v1.1 criteria

SECONDARY OUTCOMES:
Disease Control Rate | Assessed after every 4 cycles (each cycle is 14 days) for up to 24 months
  The proportion of patients who have achieved complete response (CR), partial response (PR), or stable disease (SD) following treatment initiation.
Duration of Response | Assessed after every 4 cycles (each cycle is 14 days) for up to 24 months
  Length of time from the initial detection of a measurable response (complete response or partial response) to the treatment until the first documentation of disease progression or recurrence
Progression-Free Survival | Assessed up to 24 months
  The length of time from the start of treatment until the disease progresses or the patient dies from any cause, whichever occurs first.
Overall Survival | Assessed throughout the study duration (5 years)
  Defined as the time from the start of study treatment to death due to any cause
Adverse events (Treatment-related) | Assessed throughout the study duration (5 years)
  Assessment of adverse events and their severity according to NCI CTCAE version 5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data and materials used in this study can be made available following study completion upon reasonable request to the corresponding author, subject to ethical and legal considerations and applicable data-sharing agreements.